CLINICAL TRIAL: NCT06946069
Title: Expression of CXCL11 & TEMRA in Serum of Vitiligo Patients Treated With Narrow-band UVB
Brief Title: Immunomodulatory Effects of NB-UVB and Steroids in Vitiligo: A Study on CXCL11 and TEMRA Biomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ALZAHRA MOAHMED MOHAMED ABDELHAFEZ, resident at the dermatology Surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Effects of NB-UVB and Steroids
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Vitiligo; NB-UVB
Keywords: vitiligo; NB-UVB; CXCL11; TEMRA
MeSH Terms: conditions — Vitiligo | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized controlled trial (RCT).
  Participants are randomly assigned (1:1 ratio) to one of two treatment arms:
  NB-UVB monotherapy (control group).
  NB-UVB + oral mini-pulse (OMP) steroids (intervention group).
  Both groups receive simultaneous but distinct interventions for direct comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (NB-UVB Monotherapy) (Experimental): Standard phototherapy without additional systemic treatment.
  Interventions: Radiation: NB-UVB twice weekly
- Group 2 (NB-UVB + OMP Steroids) (Experimental): Combination therapy of NB-UVB + OMP Steroids to enhance immunosuppression and repigmentation.
  Interventions: Other: NB-UVB + dexamethasone (2.5-3 mg/week)

INTERVENTIONS:
Radiation: NB-UVB twice weekly — Standard phototherapy without additional systemic treatment.
  Arms: Group 1 (NB-UVB Monotherapy)
Other: NB-UVB + dexamethasone (2.5-3 mg/week) — Combination therapy to enhance immunosuppression and repigmentation.
  Arms: Group 2 (NB-UVB + OMP Steroids)

SUMMARY:
this is a prospective, randomized controlled trial (RCT) investigating the immunological effects of narrowband UVB (NB-UVB) phototherapy-both as monotherapy and in combination with oral mini-pulse (OMP) steroids-in non-segmental vitiligo patients. The study evaluates changes in CXCL11 (a chemokine involved in T-cell recruitment) and TEMRA (terminally differentiated effector memory T cells re-expressing CD45RA) levels in serum before and after treatment.

DETAILED DESCRIPTION:
Design:

Randomized controlled trial (RCT) with two parallel arms.

Duration: Six months (including baseline and follow-up assessments).

Setting: Outpatient dermatology clinic at Assiut University Hospital, Egypt.

Objectives:

Compare the immunomodulatory effects of NB-UVB alone vs. NB-UVB + OMP steroids in vitiligo patients.

Assess CXCL11 and TEMRA levels as potential biomarkers for disease activity and treatment response.

Evaluate clinical repigmentation using Vitiligo Extent Score (VES/VESplus).

Methodology:

40 patients with stable non-segmental vitiligo will be enrolled.

20 patients will undergo serum analysis for CXCL11 and TEMRA via ELISA.

Treatment arms:

NB-UVB monotherapy (twice weekly).

NB-UVB + OMP steroids (dexamethasone 2.5-3 mg/week).

Follow-up: Clinical and immunological assessments at baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed non-segmental vitiligo (stable for ≥3 months).

Fitzpatrick skin types III-V (common in the Egyptian population).

No recent systemic therapy for vitiligo (within the last 3 months).

Exclusion Criteria:

Photosensitivity disorders (e.g., lupus, porphyria).

Pregnancy or breastfeeding.

Active infections, malignancies, or immunosuppressive conditions.

History of hypertrophic scarring or melanoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum CXCL11 & TEMRA levels | 6 months
  Measured via ELISA before and after treatment.